CLINICAL TRIAL: NCT05998070
Title: The Effect of Hip Strength Training on Upper Extremity Function and Performance in Volleyball Players
Brief Title: Effects of Hip Strengthening Training in Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Furkan Karaağaç, Physiotherapist, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7584-GOA
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Volleyball; Healthy
MeSH Terms: interventions — Sensitivity Training Groups

STUDY DESIGN:
Intervention Model Description: Hip strengthening exercises will be performed 3 times a week for 6 weeks in the exercise group. The control group will continue their routine sport training program.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Hip strengthening exercises will be performed in the training group.
  Interventions: Other: Training group
- Control group (No Intervention): The control group will continue their training and matches.

INTERVENTIONS:
Other: Training group — Hip strengthening exercises will be performed 3 times a week for 6 weeks in the training group. 3 exercises consisting of 2 sets and 10 repetitions will be performed every week. A rest interval will be given between sets.
  Arms: Training group

SUMMARY:
In order to examine the effects of hip strength training on upper extremity function and performance, 60 healthy volleyball players with an age range of 13 to 40 years will be included in our study. Shoulder joint range of motion, shoulder and hip muscle strength, upper extremity functional performance, and spike speed will be evaluated. Participants will be randomly divided into 2 groups as Training Group (TG) (will receive 6-week, 3 days a week, hip strength training in addition to their sport-specific training) and Control Group (CG) (will continue their sport-specific training).

Evaluations will be repeated 3 times before exercise training, after 6 weeks of exercise training, and at the 12th week, and the results will be analyzed.

DETAILED DESCRIPTION:
60 volleyball players will be included in our study. Assessments: 1. In the evaluation of upper extremity function and performance; strength of the shoulder internal and external rotator muscles will be measured with a hand-held dynamometer, shoulder internal and external rotation joint range of motion with a digital inclinometer, finally functional performance with closed kinetic chain upper extremity stability test and spike speed with a speed gun. 2. strength evaluation of the hip abductor, extensor, and external rotator muscles with a hand-held dynamometer. Participants will be randomly divided into 2 groups of 30 participants. The Training Group (TG) will receive 6 weeks of hip abduction, extension, and external rotation strengthening training in addition to their sport-specific training. Strengthening exercises will be done 3 days a week and every other day with a physiotherapist. Control Group (CG); will continue their sport-specific training. Evaluations will be repeated 3 times (before exercise training, after 6 weeks of exercise training, and at the end of the 12th week) and the results will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 13-40
* Volunteer to participate,
* To be training at least 2-3 session a week,
* Having played volleyball for at least 3 years, actively participating in training and competitions,
* To be able to complete all the evaluations to be made in the study

Exclusion Criteria:

* Having a systemic musculoskeletal disease,
* The occurrence of pain during the evaluations,
* History of fracture, instability or surgery in the last 6 months,
* Having an upper, lower extremity or spine injury (acute and/or active) in the last 6 months,
* Being away from sports for the last 6 months due to pain

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Shoulder strength | Baseline, 6 weeks later and 12 weeks later
  Change of shoulder internal rotation and external rotation strength(in kg, with hand held dynamometer)
Upper extremity functional performance | Baseline, 6 weeks later and 12 weeks later
  Determine the performance with Upper Extremity Closed Kinetic Chain Stabilization Test (number of touches)
Spike speed | Baseline, 6 weeks later and 12 weeks later
  Determine the performance with Spike Speed Test(in km/h, with radar gun)

SECONDARY OUTCOMES:
Shoulder range of motion | Baseline, 6 weeks later and 12 weeks later
  Change of shoulder internal and external rotation range of motion(in degree, with inclinometer)
Hip strength | Baseline, 6 weeks later and 12 weeks later
  Change of hip abduction, extension, and external rotation strength(in kg, with hand held dynamometer)

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi YESİLYAPRAK, PHD, PT, Principal Investigator — Dokuz Eylul University Department of Physiotherapy and Rehabilitation
Locations (1):
- Dokuz Eylul University Department of Physiotherapy and Rehabilitation, Izmir, Turkey (Türkiye)